CLINICAL TRIAL: NCT07093632
Title: Medium-term Results of Lower Limb Arterial Bypass
Acronym: MERLLAB
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 25-5202
Record Dates: First submitted 2025-07-29; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Peripheral Arterial Occlusive Disease; Critical Limb Ischemia; Arterial Revascularization; Arterial Bypass Surgery
Keywords: Peripheral arterial occlusive disease; critical limb ischemia; arterial revascularization; arterial bypass surgery
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Arterial Bypass Cohort: The study group consists of adult patients with symptomatic lower limb arterial disease who have undergone arterial bypass surgery.
  Interventions: Procedure: Graft dysfunction will be assessed through clinical examination and imaging follow-up to detect occlusion, pseudoaneurysm, aneurysm rupture, infection, or major amputation of the treated limb.

INTERVENTIONS:
Procedure: Graft dysfunction will be assessed through clinical examination and imaging follow-up to detect occlusion, pseudoaneurysm, aneurysm rupture, infection, or major amputation of the treated limb. — This study concerns adult subjects with symptomatic lower limb arterial disease who have undergone arterial bypass surgery and are included in the study cohort. Graft dysfunction will be assessed through clinical examination and imaging follow-up to detect occlusion, pseudoaneurysm, aneurysm rupture, infection, or major amputation of the treated limb.

SUMMARY:
Peripheral arterial occlusive disease (PAOD) is a condition affecting the arteries of the lower limbs, caused by the progressive accumulation of lipid deposits that obstruct blood vessels. At an advanced stage, PAOD may progress to critical limb ischemia (CLI), characterized by persistent pain, chronic wounds, or gangrene. This situation constitutes a medical emergency, as it may result in limb loss or threaten the life of the patient.

In this context, arterial revascularization is essential to restore adequate blood flow to the tissues. Among therapeutic options, arterial bypass surgery remains a reference strategy. The choice of bypass type, the material used (autologous vein or prosthetic graft), perioperative conditions, and clinical characteristics of patients significantly influence the success of the intervention and both short- and long-term outcomes.

When an autologous vein is not available, the use of cold-stored allogeneic vein grafts has been proposed as an alternative. Several studies have evaluated their performance, showing encouraging results in terms of graft patency and limb salvage in patients with CLI. More recently, the REVATEC study confirmed these observations in a multicenter setting in France, highlighting the feasibility and safety of this technique in routine clinical practice].

Thus, a better understanding of the factors associated with the performance of arterial bypasses and the clinical evolution of patients in real-world practice is essential to optimize management strategies.

This retrospective study aims to analyze the clinical and technical data related to arterial bypass procedures performed in patients presenting with CLI. Data will be collected at various stages of the care pathway: preoperative phase, surgical intervention, hospitalization, discharge, and 1-year follow-up. The analysis will include consecutive medical records of patients operated on between January 2018 and February 2024.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged over 18 years
* Symptomatic lower limb arterial disease
* Undergoing revascularization bypass surgery

Exclusion Criteria:

* Patients who have expressed opposition to the use of their data for research purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study concerns adult subjects with symptomatic lower limb arterial disease who have undergone arterial bypass surgery.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the incidence of arterial bypass graft dysfunction, defined by the occurrence of at least one of the following events: occlusion, pseudoaneurysm, aneurysm rupture, infection, or major amputation of the target limb. | The primary outcome will be assessed at 1-year follow-up
  The primary endpoint, graft dysfunction, will be evaluated through thorough clinical examinations combined with scheduled imaging assessments. These evaluations aim to identify any occurrence of occlusion, pseudoaneurysm formation, aneurysm rupture, infection, or major amputation of the treated limb. This comprehensive approach ensures early detection and accurate characterization of graft-related complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Louis Pradel Cardiology Hospital, Lyon, France, France